CLINICAL TRIAL: NCT05579834
Title: Perioperative Management in Terms of Hemothorax Caused by Posterior Correction
Brief Title: Hemothorax Caused by Posterior Correction Surgery for Spinal Deformity
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Cem KAYA, Asst.Prof., Gazi University
Other Study IDs: GU-260121-02
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Spinal Deformity; Hemothorax Postoperative
Keywords: spinal deformity; posterior correction surgery; hemothorax
MeSH Terms: conditions — Hemothorax

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: posterior correction surgery — Cases of hemothorax developing after posterior correction surgery for spinal deformities

SUMMARY:
Owing to the development of instruments and surgical techniques, the number of spinal deformity correction surgeries has increased significantly. The incidence of hemothorax due to posterior correction surgery for spinal deformity is reported to be as low as 0.1%, and the vast majority of these cases were treated through observation without additional intervention. However, if hemothorax that occurs is missed, it can result in increased mortality and morbidity. Furthermore, there is a paucity of data on management of hemothorax caused by posterior correction surgery. The aim of this retrospective study is to evaluate our cases of hemothorax after posterior correction surgery for spinal deformity.

DETAILED DESCRIPTION:
We retrospectively reviewed medical records of all pediatric patients who underwent posterior correction surgery from 2016 to 2021.

ELIGIBILITY:
Inclusion Criteria:

* Children who underwent posterior correction surgery for spinal deformities (age range 1-18 years)

Exclusion Criteria:

-

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children who underwent posterior correction surgery for spinal deformities (age range 1-18 years)
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-07-03 (Actual)

PRIMARY OUTCOMES:
hemothorax | 2016-2021
  hemothorax caused by posterior correction surgery for spinal deformity

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi Üniversitesi, Ankara, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided